CLINICAL TRIAL: NCT02926651
Title: Single Versus Multi-Dose Oral Tranexamic Acid in Patients at High Risk for Blood Transfusion After Total Joint Arthroplasty
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16060110
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Anemia; Arthritis; Total Knee Arthroplasty; Total Hip Arthroplasty
MeSH Terms: conditions — Anemia; Arthritis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Conventional Oral TXA, Total Hip Arthroplasty (THA) (Active Comparator): THA patients will be given three 650mg tablets of oral TXA 2 hours prior to incision with three 250mg tablets of ascorbic acid (oral TXA placebo) given 6 hours postoperatively and a final 750mg ascorbic acid dose given the morning of postoperative day 1.
  Interventions: Drug: Conventional Oral TXA (Tranexamic Acid)
- Conventional Oral TXA, Total Knee Arthroplasty (TKA) (Active Comparator): TKA patients will be given three 650mg tablets of oral TXA (Tranexamic Acid) 2 hours prior to incision with three 250mg tablets of ascorbic acid (oral TXA placebo) given 6 hours postoperatively and a final 750mg ascorbic acid dose given the morning of postoperative day 1.
  Interventions: Drug: Conventional Oral TXA (Tranexamic Acid)
- Multi-Dose Oral TXA, Total Hip Arthroplasty (THA) (Experimental): THA patients will be given three 650mg tablets of oral TXA 2 hours prior to incision with a second 1950mg oral TXA dose given 6 hours postoperatively and a final 1950mg oral TXA dose given the morning of postoperative day 1.
  Interventions: Drug: Multi-Dose Oral TXA (Tranexamic Acid)
- Multi-Dose Oral TXA, Total Knee Arthroplasty (TKA) (Experimental): TKA patients will be given three 650mg tablets of oral TXA 2 hours prior to incision with a second 1950mg oral TXA dose given 6 hours postoperatively and a final 1950mg oral TXA dose given the morning of postoperative day 1.
  Interventions: Drug: Multi-Dose Oral TXA (Tranexamic Acid)

INTERVENTIONS:
Drug: Conventional Oral TXA (Tranexamic Acid) — Three 650mg tablets of oral TXA 2 hours prior to incision with three 250mg tablets of ascorbic acid (oral TXA placebo) given 6 hours postoperatively and a final 750mg ascorbic acid dose given the morning of postoperative day 1.
  Arms: Conventional Oral TXA, Total Hip Arthroplasty (THA); Conventional Oral TXA, Total Knee Arthroplasty (TKA)
Drug: Multi-Dose Oral TXA (Tranexamic Acid) — Three 650mg tablets of oral TXA 2 hours prior to incision with a second 1950mg oral TXA dose given 6 hours postoperatively and a final 1950mg oral TXA dose given the morning of postoperative day 1.
  Arms: Multi-Dose Oral TXA, Total Hip Arthroplasty (THA); Multi-Dose Oral TXA, Total Knee Arthroplasty (TKA)

SUMMARY:
As tranexamic acid (TXA) becomes more prevalent, all patients are receiving the same dose regardless of their pre-operative risk of transfusion. Therefore the aim of the study is to determine whether or not repeated dosing of oral TXA reduces the post-operative reduction in hemoglobin, hematocrit, number of transfusions, and post-operative blood loss following primary TKA and THA surgeries in patients with low pre-operative hematocrit and high risk for transfusion. The investigators hypothesize that a multi-dose TXA regimen will significantly minimize post-operative blood loss and transfusion requirements compared to the use of a single dose regime.

DETAILED DESCRIPTION:
Total joint arthroplasty is associated with the risk of moderate to significant blood loss. Because TXA has been shown to significantly reduce the need for blood products during total joint replacement, it is now the standard of care at many institutions. Oral and intravenous TXA are equivalent, but oral TXA is cheaper and allows for ease of repeat dosing. Although low preoperative hemoglobin is a risk factor for transfusion, no studies that have compared standard TXA dosing to risk stratified dosing of TXA. The investigators hypothesize that a multi-dose TXA regimen will significantly minimize post-operative blood loss and transfusion requirements compared to the use of a single dose regimen.

At the pre-operative clinic appointment and before the day of surgery, the study staff will assess the potential subject's eligibility. Once eligibility is established, the potential subject will be approached regarding their participation in this clinical trial. The investigators will provide 48 hours before the date of surgery to allot for questions and consideration of the Informed Consent document. Once all patient questions have been answered, patients willing to be in the study will sign the Informed Consent. Patients will be randomized, via standard randomization tables that provide a 1:1 distribution of subjects between the two groups through blocked randomization, no later than the morning of surgery to either of the two treatment groups: Conventional Oral TXA Group or Multi-Dose Oral TXA Group.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* scheduled for a primary cemented TKA or cementless THA
* preoperative hematocrit less than 36%

Exclusion Criteria:

* Known allergy to TXA
* acquired disturbances of color vision
* refusal of blood products
* pre-operative use of anticoagulant therapy within five days before surgery
* a history of arterial or venous thrombotic disease (including a history of Deep Vein Thrombosis, Pulmonary Embolus, Cerebrovascular accident or Transient ischemic attack)
* pregnancy, breastfeeding
* major co-morbidities (myocardial infarction or stent placement within one year, severe pulmonary disease, renal impairment, or hepatic failure)
* undergoing a revision TKA, revision THA, hip resurfacing, or Unicompartmental Knee Arthroplasty
* younger than 18 years old
* decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients transfused | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
  Number of patients transfused per each of the 4 treatment arms
Number of units Packed Red Blood Cells (PRBCs) transfused | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
  Number of units Packed Red Blood Cells (PRBCs) transfused per each of the 4 treatment arms

SECONDARY OUTCOMES:
Post-operative reduction in hemoglobin and hematocrit | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
Calculated blood loss | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
  Based on predicted blood volume and hemoglobin balance
Cost comparison | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
  Cost differences resulted from differences in the blood transfusion rate, length of hospital stay, and management of complications as well as from the cost of the TXA itself
Complications | Post-operative and before discharge from hospital (inpatient), < 30 days from surgery
  Deep Vein Thrombosis, Pulmonary Embolus, return to the Operating Room within 30 days, superficial or deep infection, and cerebrovascular accident, transient ischemic attack or Myocardial Infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-09-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT02926651/Prot_000.pdf